CLINICAL TRIAL: NCT07019012
Title: Cofrogliptin Once Every 2 Weeks as Add-on Therapy to Metformin and Dapagliflozin Versus Daily Linagliptin in Patients With Type 2 Diabetes: A Multicenter, Randomized, Open-Label, Active-Controlled, Non-inferiority Trial
Brief Title: Cofrogliptin Once Every 2 Weeks as Add-on Therapy to Metformin and Dapagliflozin Versus Daily Linagliptin in Patients With Type 2 Diabetes.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Wuhan Central Hospital (Other); Taihe Hospital (Other); Xiangyang No.1 People's Hospital (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Xuefeng Yu, Chief of Department of Endocrinology, Tongji Hosptial Affiliated to Tongji Medical College of Huazhong University fo Science and Technology, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK7653-501
Record Dates: First submitted 2025-02-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: T2DM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cofrogliptin Add-on Group (Experimental): Triple combination therapy with cofrogliptin added to metformin and SGLT2i in type 2 diabetes mellitus (T2DM) patients who have inadequately controlled blood glucose despite adequate metformin and SGLT2i therapy for at least 12 weeks.
  Interventions: Drug: SGLT2i+Metformin+Cofrogliptin
- Linagliptin active-control Group (Active Comparator): Triple combination therapy with linagliptin as active-control drug added to metformin and SGLT2i in type 2 diabetes mellitus (T2DM) patients who have inadequately controlled blood glucose despite adequate metformin and SGLT2i therapy for at least 12 weeks.
  Interventions: Drug: SGLT2i+Metformin+Linagliptin

INTERVENTIONS:
Drug: SGLT2i+Metformin+Cofrogliptin — The combination of SGLT2i+Metformin+Cofrogliptin
  Arms: Cofrogliptin Add-on Group
Drug: SGLT2i+Metformin+Linagliptin — The combination of SGLT2i+Metformin+Linagliptin
  Arms: Linagliptin active-control Group

SUMMARY:
This study is designed to evaluate the change in glycated hemoglobin (HbA1c) levels from baseline to 24 weeks after the combination therapy of cofrogliptin, metformin and SGLT2i (dapagliflozin) in type 2 diabetes mellitus (T2DM) patients with poor control of glucose level by metformin and SGLT2i combination therapy.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the change in glycated hemoglobin (HbA1c) levels from baseline to 24 weeks after the combination therapy of cofrogliptin, metformin and SGLT2i (dapagliflozin) in type 2 diabetes mellitus (T2DM) patients with poor control of glucose level by metformin and SGLT2i combination therapy, as well as the comparison of efficacy of cofrogliptin and linagliptin. Patients will be assigned to receive the treatment of SGLT2i+metformin+cofrogliptn or SGLT2i+metformin+linagliptin.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign a written informed consent form.
* Male or female subjects aged 18 years and above .
* Meet the diagnostic criteria for Type 2 Diabetes Mellitus (T2DM).
* Have been on initial SGLT2i monotherapy (dapagliflozin) at a dose of 10 mg daily for at least 12 weeks.
* Have received metformin treatment for ≥12 weeks, with a stable dose maintained during the screening period (≥1500 mg/day if tolerable or at the maximum tolerated dose (<1500 mg/day but ≥1000 mg/day), and no dosage adjustment).
* HbA1c levels within the range: 7.0% < HbA1c ≤ 10.0%.
* Fasting plasma glucose (FPG) < 15 mmol/L.
* Body Mass Index (BMI) ≤ 40 kg/m2.
* Estimated Glomerular Filtration Rate (eGFR) ≥ 60 ml/min/1.73m2.
* Agree to maintain the same diet and exercise habits throughout the trial period, willing and able to accurately use a home blood glucose meter for self-monitoring of blood glucose (SMBG) and keep records.

Exclusion Criteria:

* Type 1 Diabetes Mellitus.
* Any type of secondary diabetes.
* Pending or having undergone pancreatic or β-cell transplantation.
* History of pancreatitis or pancreatic resection.
* Complicated with diabetic ketoacidosis or hyperosmolar coma.
* Moderate or severe hepatic insufficiency of any cause. Hepatic insufficiency is defined as screening period levels of ALT (SGPT), AST (SGOT), or alkaline phosphatase serum levels exceeding 3 times the upper limit of normal (ULN).
* Acute coronary syndrome (ST-elevation myocardial infarction, non-ST-elevation myocardial infarction, unstable angina), stroke, or transient ischemic attack (TIA) within the last 3 months.
* Uncontrolled hypertension: systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg.
* Hemoglobin levels < 10 g/l or 100 mg/dl.
* More than 2 recurrent genitourinary infections within the last 3 months.
* History of bariatric surgery or other gastrointestinal surgeries leading to chronic malabsorption within the last 2 years.
* Weight instability due to anti-obesity medication within the last 3 months or any other treatment (such as surgery, aggressive diet plans) at screening.
* History of cancer (excluding basal cell carcinoma) and/or cancer treatment within the last 5 years.
* Human Immunodeficiency Virus (HIV) infection.
* Severe peripheral vascular disease.
* Hematological malignancy or any disorder causing hemolysis or erythrocyte instability (e.g., malaria, babesiosis, hemolytic anemia).
* Concurrent immune system diseases or currently receiving systemic corticosteroid therapy.
* Changes in thyroid hormone dosage within the last 6 weeks, or any other uncontrolled endocrine or metabolic disorder outside of T2DM.
* Alcohol or drug abuse within the last 3 months that may reduce trial compliance, or any chronic condition deemed by the investigator as likely to reduce study compliance or medication adherence.
* Known allergy to the trial medication components or other chemically similar drugs or excipients.
* Pregnant women, women planning pregnancy during the study or breastfeeding, subjects unwilling to use reliable contraception (including condoms, spermicides, or intrauterine devices) from signing the informed consent form until 28 days after the last dose of trial medication, or women planning to use progesterone-containing contraceptives during this period. Men with plans for conception during the study.
* Participation in any other clinical study within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The change in glycated hemoglobin (HbA1c) levels | From enrollment to the end of treatment at 24 weeks
  To evaluate the change in glycated hemoglobin (HbA1c) levels from baseline to week 24 after triple combination therapy with cofrogliptin added to metformin and sodium-glucose cotransporter 2 inhibitor(SGLT2i) in type 2 diabetes mellitus (T2DM) patients who have inadequately controlled blood glucose despite adequate metformin and SGLT2i therapy.

SECONDARY OUTCOMES:
HbA1c target rate | From enrollment to the end of treatment at 24 weeks
  Proportion of subjects achieving HbA1c < 7.0% and < 6.5% at 24 weeks.
2h-PPG and FPG | From enrollment to the end of treatment at 24 weeks
  Changes in 2-hour postprandial plasma glucose (2h-PPG) and fasting plasma glucose (FPG) from baseline at 12 and 24 weeks.
Change in HbA1c levels | From enrollment to the end of treatment at 24 weeks
  Change in HbA1c levels from baseline at 24 weeks.
Weight related items | From enrollment to the end of treatment at 24 weeks
  Changes in body weight, fasting C-peptide, HOMA-IR, and HOMA-β from baseline at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: XueFeng Yu, Doctor, Principal Investigator — Tongji Hosptial Affiliated to Tongji Medical College of Huazhong University fo Science and Technology
Locations (1):
- Wuhan University People's Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Scientific data should be analyzed before release